CLINICAL TRIAL: NCT04299646
Title: A Phase II Study Assessing Stereotactic Radiotherapy in Therapeutic Strategy of Oligoprogressive Renal Cell Carcinoma Metastases
Acronym: GETUG-StORM-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government); GETUG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-StORM-01
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Renal Cell Carcinoma; Radiotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Non randomized phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steretactic radiotherapy plus systemic treatment (Experimental)
  Interventions: Radiation: Steretactic radiotherapy

INTERVENTIONS:
Radiation: Steretactic radiotherapy — Steretactic radiotherapy

SUMMARY:
Every year, 12500 primary renal cell carcinoma (RCC) are diagnosed in France. Metastases occur in half of RCC patients.

Management of metastatic RCC is based on systemic treatments (targeted therapies/immunotherapy). However, resistance to systemic treatment is frequent. In case of progression, usual therapeutic attitude is initiating another systemic therapy.

Because of the emergence of resistant tumor clonal cells, some patients progress only on few sites while the rest of tumor burden is controlled. In this setting named oligoprogressive disease [isolated progression of <3-5 metastase(s)], ablative treatments of these evolving metastatic sites could allow a disease control and a reduced risk of new metastases occurrence by tumor-cell reembolization. Such strategy is challenging to prolong ongoing systemic treatment and delay further lines.

Although RCC was considered radioresistant and radiotherapy with conventional fractionation was mainly used for palliation of symptoms, stereotactic radiotherapy (SRT), by delivering high dose in one or few fractions, allows local control for about 90% of RCC metastases through various radiobiological pathways. Furthermore, some data suggest that high-dose focal irradiation of RCC could induce a systemic antitumor response mediated by immunologic effectors(1). This phenomenon ("abscopal effect") could be enhanced in patients under immunotherapy, including anti-PD1.

Several retrospective studies and one non-randomized phase-II study highly suggest the interest of SRT as focal ablative treatment in RCC oligometastases with excellent local control rates and low toxicity(2,3).

Furthermore, the multicentric retrospective study the sponsor recently conducted within the GETUG group among 101 metastatic RCC patients with oligoprogression under systemic therapy highlighted that SRT on progressive sites provided a median of 8.6-month progression-free survival and allowed to continue current systemic line for 10.5 months.

However, to date, there are no prospective data assessing the interest of SRT for management of oligoprogressive metastatic RCC.

The sponsor aim to prospectively evaluate the interest of SRT as a therapeutic strategy for local control of oligoprogressive metastatic RCC under ongoing systemic treatment, and consequently delay subsequent systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clear cell renal cancer histologically proved (association with other histologic component are permitted)
* Patients of good or intermediate prognostic, according to Heng criteria
* Extracerebral metastatic disease documented with imagery
* Patients treated in first or second line systemic therapy
* Systemic treatment may be targeted therapies (tyrosine kinase inhibitors or mammalian target of rapamycin inhibitors) and/or immunotherapy according to French applicable standards; patients treated in a clinical trial are also eligible if allowed by trial sponsor
* Oligoprogressive disease documented with imagery, defined as the emergence or progression of 1 to 3 metastases and progression localized in up to 2 organs
* Oligoprogressive disease confirmed with 2 CT scans performed 2 months apart
* At least one measurable progressing metastasis according to R.E.C.I.S.T. criteria v1.1
* All oligoprogressive target lesions measuring ≤ 4 cm
* Good general condition (WHO performance status ≤ 2)
* All progressive lesions have to be accessible to SRT, performed concurrently or sequentially
* No contraindication to systemic therapy and stereotactic radiation therapy
* Patients aged 18 years or older
* Signed informed consent form
* Patients affiliated to the social security system

Exclusion Criteria:

* More than 3 progressive metastases
* Non measurable disease according R.E.C.I.S.T. criteria
* Patients who received 3 or more lines of systemic therapy
* Inability to treat all progressive metastatic sites with SRT
* Previous radiation therapy performed in ≥ 1 target lesion
* At least 1 oligoprogressive target lesion measuring > 4 cm
* Presence of brain metastases
* Presence of ultra-central pulmonary metastasis
* Progressing metastasis in a long bone
* At least 1 progressive metastasis requiring surgical treatment
* Current or past history of second neoplasm diagnosed within the last 5 years
* Pregnancy or breast feeding or inadequate contraceptive measures
* Patients who cannot be adequately followed up
* Patient deprived of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months post-randomization

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Until 1 month after end of treatment
Local control rate | 3, 6 and 12 months after randomization
Overall control rate | 3, 6 and 12 months after randomization

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - Clinique Claude Bernard, Albi
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - Radiothérapie Bordeaux Nord Aquitaine, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - Centre Georges François LECLERC, Dijon
  - Institut de cancérologie de Bourgogne (Dijon, Auxerre, Chalon sur Saône), Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Centre de radiothérapie Guillaume le Conquérant, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - Institut Paoli Calmette, Marseille
  - CHR, Metz
  - ICM, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Haute Energie, Nice
  - Institut Curie, Paris
  - Groupement de radiothérapie Oncologie des Pyrénées, Pau
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Etienne
  - Polyclinique de l'Ormeau, Tarbes
  - IUCT, Toulouse
  - Centre marie Curie, Valence
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No